CLINICAL TRIAL: NCT01355237
Title: Use and Effectiveness of a Model Integrative Care Clinic in an Academic Hospital: Study II - Observational Cohort Study of Chronic Low Back Pain
Brief Title: Observational Cohort Study of Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Julie E. Buring, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 1R01AT005065-01A1-2; 1R01AT005065-01A1 (NIH)
Record Dates: First submitted 2011-05-12; First posted 2011-05-18 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Back Pain Lower Back Chronic
Keywords: Complementary and alternative medicine (CAM)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- OCC Patients: Patients being treated for chronic low back pain at the Osher Clinical Center of Brigham and Women's Hospital
- Comparison: Patients being treated for chronic low back pain at Brigham and Women's Hospital, other than at Osher Clinical Center

SUMMARY:
This research study is being done to understand the outcomes of back pain treatment and costs associated with it in an academic hospital outpatient setting. The investigators will conduct a prospective observational cohort study to assess the clinical outcomes and utilization of health care services of 175 Osher Clinical Center (OCC) patients with chronic low back pain (CLBP) compared with a comparison group of 175 non-OCC CLBP patients treated within Brigham and Women's Hospital. Outcomes will include assessment of functional status, symptom relief, satisfaction with care, health-related quality of life, and worker productivity, and will be measured in person at baseline, and by phone by an interviewer blinded to cohort group at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 3 months or more of chronic low back pain or 6 months or more of intermittent low back pain OR
* having at least one of a list of ICD-9 diagnostic codes for uncomplicated low back pain
* having two or more visits for back pain within the past two years; one of these visits must have happened within the past year (as a screening marker of chronicity)

Exclusion Criteria:

* under the age of 21
* unable to understand English
* have complicated low back pain (e.g. history of back pain related to cancer, fracture, or infection)
* unable to participate in the phone follow-up for the next one-year period.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The CLBP patients will be identified from two different sources at Brigham and Women's Hospital (BWH): those coming to be treated at the OCC, and those coming to non-OCC physician providers at BWH (comparison group).
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2012-02; Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in functional disability related to low back pain | 6 months
  Measured by change in Modified Roland Morris disability scale (0-23 points)
Change in Bothersomeness of pain | 6 months
  Measured by change in bothersomeness scale (On a scale of 0-10)

SECONDARY OUTCOMES:
Cost-effectiveness of integrative care for chronic low back pain | 12 months
  Measured by utilization of health care services and productivity in the workplace

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Buring, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States